CLINICAL TRIAL: NCT06181266
Title: A Phase 1/1b Study Evaluating the Safety, Pharmacology, and Clinical Effect of ZH9 Treatment in Patients With Non-Muscle Invasive Bladder Cancer
Brief Title: A Phase 1/1b Study of ZH9 Treatment in Patients With Non-Muscle Invasive Bladder Cancer
Acronym: PARADIGM-1
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Prokarium Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRK-23101
Record Dates: First submitted 2023-12-12; First posted 2023-12-26 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: NMIBC; High Risk NMIBC; Non Muscle Invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: In Part 1, the safety, tolerability, and pharmacology of ZH9 administered as an IVI will be evaluated in a single ascending dose cohort in patients with NMIBC. Part 1 may examine up to 4 dose levels.
  In Part 2, the safety, tolerability, and pharmacology of ZH9 oral prime followed by ZH9 IVI will be evaluated in 2 cohorts in patients with NMIBC at the doses and schedule established in Part 1.
  In Part 3, the safety, pharmacology, and clinical efficacy of ZH9 (oral prime and IVI) will be further evaluated in 2 expansion cohorts of patients with recurrent intermediate- and high-risk NMIBC.
Masking Description: All administrations of ZH9 as an IVI will be open-label in Parts 1, 2, and 3. In Part 2 only, patients will be randomized 1:1 to receive either ZH9 or placebo oral prime. The oral priming condition will be conducted in a double-blind, placebo-controlled manner. The randomization list will only be made available to the unblinded pharmacist dispensing the study drug. At each clinical site, an unblinded pharmacist will be assigned to prepare the blinded study drug for administration (ZH9 oral prime or placebo).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Level 1 - ZH9 (Experimental): Part 1 will evaluate SAD of ZH9 administered as an IVI in patients with recurrent NMIBC. A standard 3+3 escalation design will be employed with the dose levels
  Interventions: Drug: ZH9
- Dose Level 2 - ZH9 (Experimental): Part 1 will evaluate SAD of ZH9 administered as an IVI in patients with recurrent NMIBC. A standard 3+3 escalation design will be employed with the dose levels
  Interventions: Drug: ZH9
- Dose Level 3 - ZH9 (Experimental): Part 1 will evaluate SAD of ZH9 administered as an IVI in patients with recurrent NMIBC. A standard 3+3 escalation design will be employed with the dose levels
  Interventions: Drug: ZH9
- Dose Level 4 - ZH9 (Experimental): Part 1 will evaluate SAD of ZH9 administered as an IVI in patients with recurrent NMIBC. A standard 3+3 escalation design will be employed with the dose levels
  Interventions: Drug: ZH9

INTERVENTIONS:
Drug: ZH9 — ZH9 is a live attenuated S. enterica serovar Typhi ZH9 [Ty2 ΔaroC ΔssaV]), a differentiated novel microbial immunotherapy.

SUMMARY:
This is a first-in-human, multicenter, Phase 1/1b, 3-part, double-blind study of ZH9 in patients with recurrent NMIBC who are eligible for intravesical therapy. In Part 1, the safety, tolerability, and pharmacology of ZH9 IVI will be evaluated in a single ascending dose (SAD) patient cohort. In Part 2, the safety, tolerability, and pharmacology of ZH9 oral prime followed by ZH9 IVI will be evaluated in 2 patient cohorts at the doses and schedule established in Part 1. In Part 3, the safety, pharmacology, and clinical efficacy of ZH9 will be further evaluated in 2 expansion cohorts of patients with recurrent intermediate- and high-risk NMIBC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically documented recurrence of NMIBC
* BCG unresponsive (BCG naïve patients may be enrolled if they have received at least 1 line of adequate intravesical standard of care (SOC) treatment and are either not candidates for BCG or do not have access to BCG (e.g., BCG shortage))
* Eastern Cooperative Oncology Group Performance Status 0-1
* Adequate organ and marrow function
* Highly effective contraception if risk of conception exists.
* A female participant is eligible if not pregnant, not breastfeeding, not a woman of childbearing potential (WOCBP) or is a WOCBP that uses highly effective contraception.

Exclusion Criteria:

* Received treatment with any local or systemic antineoplastic therapy within 3 weeks or 5× the plasma half-life prior to first dose of ZH9
* Major surgery or radiation within the 3 weeks prior to Screening (TURBT is not considered major surgery)
* Concurrent urinary tract infection or history of clinically significant polyuria
* Symptoms consistent with typhoid
* Evidence of infection within 2 weeks of the first dose of ZH9
* Significant 12-lead electrocardiogram abnormalities
* History of malignancy within the previous 12 months
* History of allogeneic tissue/solid organ transplant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities | 28 days
  Toxicity will be evaluated according to the NCI CTCAE Version 5.0

SECONDARY OUTCOMES:
Rate of complete pathologic response | 3, 6, and 12 months
  Rate of complete pathologic response at determined timepoints by cystoscopy, urine cytology, and if needed for pathological confirmation, biopsy
Rate of recurrence-free survival and duration or response | 3, 6, and 12 months
  Rate of recurrence-free survival and duration of response as determined by cystoscopy and urine cytology
Rate of CR | 6 and 12 months
  Rate of CR as determined by biopsy in patients with CIS at baseline
Proportion of patients with cystectomy-free survival | 6 and 12 months
  Proportion of patients with cystectomy-free survival as determined by cystoscopy and urine cytology
Rate of progression-free survival | 12 months
  Rate of progression-free survival, including disease progression and all-cause death
Overall response rate and recurrence-free rate | 6 and 12 months
  Overall response rate and recurrence-free rate in the bladder following IVI
Change from baseline in systemic and local inflammatory markers in the bladder | 12 months
  Change from baseline in systemic and local inflammatory markers in the bladder as defined by clinical laboratory safety assessments (serum chemistry, hematology, urinalysis)

CONTACTS AND LOCATIONS:
Overall Officials: Josefin-Beate Holz, MD, Study Director — Prokarium Ltd
Locations (4):
- United States (4):
  - Michael G. Oefelein Clinical Trials, Bakersfield, California
  - Duke Health-Duke Cancer Center, Durham, North Carolina
  - Carolina Urologic Research Center, LLC, Myrtle Beach, South Carolina
  - Urology San Antonio Medical Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided